CLINICAL TRIAL: NCT06338514
Title: The Effectiveness of Dry Needling Treatment in Patients Diagnosed With Dorsalgia Accompanied by Myofascial Pain Syndrome.
Brief Title: The Effectiveness of Dry Needling Treatment in Patients Diagnosed With Dorsal Myofascial Pain Syndrome.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Hasan Hüseyin Gökpınar, Assistant Professor, Kutahya Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KutahyaHSU-DRYNEEDLE-dorsalgia
Record Dates: First submitted 2024-03-24; First posted 2024-03-29 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Myofascial Trigger Point Pain
MeSH Terms: conditions — Myofascial Pain Syndromes

STUDY DESIGN:
Intervention Model Description: A two-group, sham-controlled, double-blind, prospective, randomized controlled trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: In the dry needling application, patients will be blinded to the groups they are randomized into. The evaluator will also be unaware of which group the patients belong to. The practitioner will perform the procedures in both groups using ultrasound guidance, targeting the standard trigger points in the painful dorsal trapezius and rhomboid muscles in the study group, and targeting subcutaneous fatty tissue in the same regions in the sham group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dry needling group (study group) (Active Comparator): Real dry needling into the muscle under ultrasound guidance.
  Interventions: Other: Real dry needling
- Sham dry needling group (control group) (Sham Comparator): Sham dry needling into the subcutaneous fatty tissue under ultrasound guidance.
  Interventions: Other: Sham dry needling

INTERVENTIONS:
Other: Real dry needling — dry needling into the muscle under ultrasound guidance.
  Arms: Dry needling group (study group)
Other: Sham dry needling — dry needling into the subcutaneous fatty tissue under ultrasound guidance.
  Arms: Sham dry needling group (control group)

SUMMARY:
Back pain is commonly seen in the working-age population, with the peak occurrence around the age of 40. Its frequency does not increase with age and is not associated with age-related degenerative changes in the spine. Especially when the underlying cause is conditions such as myofascial pain syndrome (MPS), where regional muscle sensitivity in the rhomboid and trapezius areas is prominent, dry needling treatment has become increasingly popular and the subject of numerous studies in recent years. In the diagnosis of MPS, two valuable findings include the detection of a taut band upon palpation and the presence of trigger points in muscle fibers with mild finger pressure. The study we are planning involves a double-blind efficacy trial where real and sham dry needling procedures will be performed under ultrasound guidance, ensuring that both the patient and the evaluator are blinded. This study design has the potential to make a significant contribution to the literature in this field.

DETAILED DESCRIPTION:
The study aims to enroll 60 patients aged between 18 and 80 years who present to the Physical Therapy and Rehabilitation Clinic of KSBÜ Evliya Çelebi Training and Research Hospital with complaints of dorsalgia and clinically diagnosed with Dorsal Myofascial Pain Syndrome. After signing informed consent forms, eligible patients will be randomized into two different groups using a random number table (randomizer.org) according to inclusion and exclusion criteria. This study will be a two-group, sham-controlled, double-blind, prospective, randomized controlled trial. Patients and the evaluator will be blinded to group allocation, with only the physician administering the dry needling treatment being aware of the assignment.

In the dry needling application, thinner needles with a gauge of 27 and a length of 5 cm, which are significantly finer than conventional standard injection needles, will be used in both the study and sham groups. These needles minimize tissue irritation due to their finer tip, targeting the trigger points in the trapezius and rhomboid muscles on the standard painful side in the study group and the subcutaneous fatty tissue in the same regions in the sham group.

Throughout the study period, all patients in both groups will be instructed in detail on the daily exercises they need to perform (trapezius stretching and rhomboid stretching exercises), as well as on important considerations (avoiding prolonged static positions, etc.). They will be encouraged to perform these exercises daily and mark their completion. Additionally, they will be informed about the selection and usage of medications (only paracetamol) that they can use when necessary, along with instructions on adherence and marking on the provided follow-up form. The entire process will be monitored weekly through the follow-up form provided to the patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed with Dorsal Myofascial Pain Syndrome associated with rhomboid and trapezius trigger point.
* Having a shoulder pain Visual Analog Scale (VAS) score of 6 or higher.
* Ability to read and write

Exclusion Criteria:

* History of spinal surgery.
* Lesions, atrophy, or scars in the skin around the back.
* Undergoing physiotherapy targeting the back and lumbar region in the last 6 months.
* Undergoing an interventional procedure for back or lumbar pain in the last 3 months.
* Use of steroids in the last 1 month.
* Special conditions such as epilepsy, pregnancy, injection phobia, etc.
* Inability to comply with the restriction on the use of steroid and non-steroidal anti-inflammatory drugs during the treatment period.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-04-25 (Actual); Primary Completion 2025-10-10 (Estimated); Study Completion 2025-11-10 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | [Time Frame: Time frame 1: Up to 24 hour before the first intervention, Time frame 2: Up to 24 hour before the second intervention, Time frame 3: One week after the last intervention, Time frame 4: One month after the last intervention]
  "Visual Analog Scale (VAS)" is a measurement instrument often used in healthcare to assess the intensity or characteristics of subjective experiences such as pain. It typically consists of a straight line, usually 10 centimeters in length, with endpoints representing extremes (e.g., "no pain" to "worst imaginable pain"). Patients mark on the line to indicate their subjective experience, and the distance from one endpoint provides a numerical score representing the intensity of the sensation being measured. The VAS is commonly employed in pain assessment but can also be adapted for various other subjective evaluations.
Patient-Specific Functional Scale | [Time Frame: Time frame 1: Up to 24 hour before the first intervention, Time frame 2: Up to 24 hour before the second intervention, Time frame 3: One week after the last intervention, Time frame 4: One month after the last intervention]
  "Patient-Specific Functional Scale" (PSFS). The PSFS is a self-report outcome measure commonly used in healthcare, particularly in physical therapy and rehabilitation settings. It is designed to assess the patient's perceived difficulty in performing specific activities that are relevant to their daily life and function. Identification of Activities: The patient is asked to identify and list three to five activities that they find challenging or have difficulty performing due to their condition or symptoms. Rating Scale: For each identified activity, the patient is asked to rate their current level of difficulty on a numerical scale, often ranging from 0 to 10. A score of 0 indicates no difficulty, while 10 indicates the maximum difficulty. Follow-up Assessments: The same activities and rating scale are used in follow-up assessments to track changes over time or in response to interventions.
Pressure Pain Threshold Measurement | [Time Frame: Time frame 1: Up to 24 hour before the first intervention, Time frame 2: Up to 24 hour before the second intervention, Time frame 3: One week after the last intervention, Time frame 4: One month after the last intervention
  "Pressure Pain Threshold Measurement" refers to the assessment of the amount of pressure applied to a specific point on the body before the individual perceives it as painful. This measurement is commonly used in clinical settings to evaluate pain sensitivity and threshold. The process involves gradually applying pressure to a specific area until the individual signals that they begin to feel pain. It is a quantitative way to assess pain perception and is often utilized in research, physical therapy, and other healthcare disciplines to understand pain levels and responses.

SECONDARY OUTCOMES:
What does Oswestry stand for? The Oswestry Disability Index (ODI) | [Time Frame: Time frame 1: Up to 24 hour before the first intervention, Time frame 2: One week after the last intervention, Time frame 3: One month after the last intervention]
  What does Oswestry stand for? The Oswestry Disability Index (ODI) is a common questionnaire used to evaluate functional outcomes and physical functioning in patients with acute or chronic low back pain. This questionnaire yields a subjective percentage score that grades the level of physical function or disability. Each section is scored on a 0-5 scale, 5 representing the greatest disability. The index is calculated by dividing the summed score by the total possible score, which is then multiplied by 100 and expressed as a percentage. Thus, for every question not answered, the denominator is reduced by 5. The Oswestry Disability Index (ODI) is calculated based on each score of the ODQ, which consists of ten items. Each of the ten items is scored from 0 to 5, and the total is added and multiplied by 2. Therefore, the ODI ranges from 0 to 100. A higher score on the ODI indicates a more severe disability caused by LBP.
The 12-item Short-Form Health Survey version 2 (SF-12v2) | [Time Frame: Time frame 1: Up to 24 hour before the first intervention, Time frame 2: One week after the last intervention, Time frame 3: One month after the last intervention]
  The SF-12v2 is a health-related quality-of-life questionnaire consisting of twelve questions that measure eight health domains to assess physical and mental health. Physical health-related domains include General Health (GH), Physical Functioning (PF), Role Physical (RP), and Body Pain (BP). What is the maximum score for SF-12? Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning

CONTACTS AND LOCATIONS:
Overall Officials: Hasan H Gökpınar, Ass. Prof., Principal Investigator — Kutahya Health Sciences University
Locations (1):
- Kütahya Health Sciences University, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No